CLINICAL TRIAL: NCT02584673
Title: Computer Assisted Instrument Guidance (CAIG) For Arterial Line Placement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clear Guide Medical (Industry)
Collaborators: The Cooper Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CGM 15-001
Record Dates: First submitted 2015-10-21; First posted 2015-10-22 (Estimated); Results first posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-05

CONDITIONS: Arterial and Midline Catheterization

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- CAIG (Experimental): The participants in this group (test group) will utilize the same procedure utilizing existing ultrasound equipment with the supplemental CAIG system.
  Interventions: Device: Computer Assisted Instrument Guidance (CAIG), which supplements existing ultrasound capabilities.
- Control (No Intervention): The participants in the control group will receive the procedure with traditional ultrasound methods and equipment.

INTERVENTIONS:
Device: Computer Assisted Instrument Guidance (CAIG), which supplements existing ultrasound capabilities. — The Clear Guide ONE is a Computer Assisted Instrument Guidance (CAIG) device which supplements existing ultrasound capabilities. The participants randomly selected (out of 100 patients) for use of the Clear Guide ONE (test group) will receive ultrasound guidance as well as CAIG from the MDs performing the procedure.
  Other Names: Clear Guide ONE
  Arms: CAIG

SUMMARY:
The objective of this research is to verify the procedural improvements enabled by use of a CAIG system to supplement existing ultrasound guided, needle-based procedures. The primary focus will be procedures performed by the Anesthesia department.

DETAILED DESCRIPTION:
The study will utilize two groups of patients: control and test. The control group will receive the procedure with traditional methods and equipment currently in use at Cooper University. The test group will receive the same procedure utilizing existing ultrasound equipment with the supplemental CAIG system. It is anticipated that 100 patients will be included in the study. After each procedure completion times, number of needle repositions, and punctures will be recorded along with an "ease of procedure" self-reported qualitative metric from the physician performing the procedure.

ELIGIBILITY:
Inclusion Criteria:

* Undergoing vessel catheterization
* Able to give written informed consent

Exclusion Criteria:

* Unable to give informed consent
* Prisoners, pregnant women, and children

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12-09 (Actual); Study Completion 2016-12-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Irwin Gratz, DO, Principal Investigator — The Cooper Health System
Locations (1):
- The Cooper Health System, Camden, New Jersey, United States

REFERENCES:
- [Derived] Flumignan RL, Trevisani VF, Lopes RD, Baptista-Silva JC, Flumignan CD, Nakano LC. Ultrasound guidance for arterial (other than femoral) catheterisation in adults. Cochrane Database Syst Rev. 2021 Oct 12;10(10):CD013585. doi: 10.1002/14651858.CD013585.pub2. PMID 34637140

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | CAIG | Control
Started | 15 | 15
Completed | 15 | 15
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CAIG | Control | Total
Number analyzed (Participants) | 15 | 15 | 30
Age, Customized [Count of Participants; unit: Participants] — At least 18 years of age Population: This data was not collected
Sex/Gender, Customized [Count of Participants; unit: Participants] | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 15 | 15 | 30

OUTCOME MEASURES:

1. Primary Outcome: Time Needed to Correctly Insert the Arterial or Midline Catheter.
Time Frame: Immediately following intervention (within 2 hours)
Measure: Mean (Standard Deviation); unit: Seconds
Arm/Group | CAIG | Control
Number analyzed (Participants) | 15 | 15
Seconds | 30.07 (28.63) | 44.76 (33.96)

2. Secondary Outcome: Clinician Rating of the Device
Time Frame: Immediately following intervention (within 2 hours)
Population: This data was not collected
Arm/Group | CAIG | Control
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Number of Attempts
Description: Number of instrument pricks before target is reached
Time Frame: Immediately following intervention (within 2 hours)
Population: This data was not collected
Arm/Group | CAIG | Control
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Number of Times Needle Needs Repositioning
Time Frame: Immediately following intervention (within 2 hours)
Population: This data was not collected
Arm/Group | CAIG | Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | CAIG | Control
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 0/15 | 0/15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No